CLINICAL TRIAL: NCT06084806
Title: Test-retest Evaluation of [18F]F-AraG PET in Non-small Cell Lung Cancer (NSCLC) Patients
Brief Title: Test-retest Evaluation of [18F]F-AraG PET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CellSight Technologies, Inc. (Industry)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CST-FARAG-IO-UIOW-201-TRT
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Advanced non small cell lung cancer (NSCLC) patients (Experimental): Patients will undergo two [18F]F AraG PET/CT scans within 7 days of each other prior to receiving treatment
  Interventions: Drug: [18F]F-ARAG PET

INTERVENTIONS:
Drug: [18F]F-ARAG PET — Two imaging sessions

SUMMARY:
This pilot study aims to evaluate the test-retest variability of [18F]F-AraG-PET imaging in patients with advanced NSCLC tumors. The main objectives of the study are to quantify the uptake of [18F]F-AraG in tumors and lymphoid tissue in two consecutive scans spaced not longer than 7 days apart from each other to estimate the magnitude of physiologic and measurement variability. To explore these objectives, eligible subjects will undergo two [18F]F-AraG PET/CT scans within 7 days of each other prior to receiving treatment. This study is a single-site, open-label, non-randomized, single-arm pilot trial. Patients and care providers will not be blinded to any part of the study.

DETAILED DESCRIPTION:
Checkpoint inhibitor therapy has led to impressive clinical successes, providing objective and durable responses in patients with advanced cancers that previously had very few treatment options. Unfortunately, immunotherapy works only in a relatively small fraction of patients with solid tumors.

The current standard of care anatomic imaging adequately assessed treatment efficacy in the pre-immunotherapy era, when tumor volume burden directly correlated with clinical outcomes. However, anatomic imaging is found to be limited due to the cellular and molecular nature of early responses to immunotherapy. PET imaging is a sensitive technique that uses radiolabeled agents to visualize the distribution of specific molecular targets in the body. Based on its ability to pinpoint molecular activity, PET imaging agents that target key players of the immune response could offer a powerful noninvasive tool for evaluation of complex immunologic processes within the body.

[18F]F-AraG was developed as an agent for imaging activated T cells (Namavari et al., 2011)). [18F]F-AraG is a 18F-labeled analog of 9-b-D-Arabinofuranosylguanine a compound that has shown selective accumulation in T cells (Eriksson, et al., 1994) and whose prodrug, nelarabine, is FDA-approved for treatment of patients with T cell acute lymphoblastic leukemia and T cell lymphoblastic lymphoma. [18F]F-AraG is independent of the type of immunotherapy regimen being administered adoptive cell therapy, checkpoint inhibitors, cancer vaccines or a combination of immunotherapy and conventional medicines. In vivo, real time imaging of activated T cells in solid tumors before and at a timepoint during and after CkIT therapy can help understand the effects of checkpoint blockade therapy. Repeatability, as an estimate of the magnitude of change that distinguishes normal physiologic and measurement variability from true biologic change, is important to interpreting changes encountered on PET scans in the response-to-treatment setting.

This study will establish test-retest variability of [18F]F-AraG uptake in tumors (primary and metastatic sites) and lymphoid tissue in NSCLC patients prior to start of therapy. The results lead to a better understanding of the parameters affecting signal quantitation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (>18 years old) with a histologically confirmed NSCLC and a candidate to receive immunotherapy as monotherapy or as combination therapy for advanced/metastatic disease.
2. Measurable disease.
3. ECOG performance status of 0, 1 or 2.

Exclusion Criteria:

1. Serious comorbidities that in the opinion of the investigator/sponsor could compromise protocol objectives.
2. Pregnant women or nursing mothers.
3. Patients with severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
[18F]F-AraG Test - Re Test | 7 days
  • Quantitative assessment of tracer uptake by Standardized Uptake Value (SUV) based measurements within volumes of interest on two consecutive [18F]F AraG PET scans

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Furqan, M.D., Principal Investigator — Holden Comprehensive Cancer Center
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided